CLINICAL TRIAL: NCT01597349
Title: An Exploratory, Randomized, Placebo Controlled, Double Blind, Parallel Arm Dose Ranging Study to Determine the Antitussive Effects of FP01 Lozenges in Subjects With Cough Due to Upper Respiratory Tract Infection
Brief Title: Antitussive Effects of FP01 Lozenges in Subjects With Cough Due to Upper Respiratory Tract Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN01-002-A
Record Dates: First submitted 2012-05-09; First posted 2012-05-14 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Acute Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- FP01 High dose (Experimental)
  Interventions: Drug: FP01
- FP01 Low dose (Experimental)
  Interventions: Drug: FP01
- Placebo (Placebo Comparator)
  Interventions: Drug: FP01

INTERVENTIONS:
Drug: FP01 — Lozenge 3 times per day, low dose, high dose, or placebo for 48 hours.

SUMMARY:
The purpose of this research study is to learn how effective and safe FP01 lozenges are when given to subjects with a cough due to an upper respiratory tract infection. The study will include subjects who have an upper respiratory tract infection, with a cough of less than six weeks duration.

ELIGIBILITY:
gastroesophageal INCLUSION CRITERIA

1. Subject must state that they have had a "cold" for < 14 days. A "cold" is defined as:

   * Moderate or severe rhinorrhea (i.e., using 2 or more tissues per hour for any 1 hour within 12 hours preceding study screening AND
   * At least one other respiratory symptom (cough, pharyngeal symptoms [sore throat], nasal congestion of moderate or severe intensity, headache, etc.)
2. Subject must exceed a cough severity threshold (VAS) during screening visit (Cough Severity VAS score ≥ 40 mm).
3. Subjects who recall that their average number of days with cough during their usual cold history is 3 or greater (URTI cough history > 3).
4. Subjects who do not smoke or use nicotine or nicotine containing products. Ex-smokers/ex-tobacco users must have stopped using tobacco products for at least 6 months prior to study screening.
5. Female subjects should be either post-menopausal (amenorrhea for at least 12 consecutive months), surgically sterile, or women of child-bearing potential (WOCP) with a negative serum beta human chorionic gonadotropin (HCG) pregnancy test prior to entering the study and who are using or agree to use an acceptable method of contraception as determined by the Investigator. Acceptable contraceptives include abstinence OR intrauterine devices (IUDs), hormonal contraceptives (oral, depot, patch or injectable) for ≥ three months prior to screening OR use of double barrier methods such as condoms or diaphragms with spermicidal gel or foam.
6. Subject must sign an Institutional Review Board approved informed consent and agree to complete required clinic visits.

EXCLUSION CRITERIA

1. Subject who are using antibiotics at study screening or for whom antibiotics are currently indicated as determined by the Investigator.
2. History of cough of greater than 6 weeks in duration.
3. History of any chronic pulmonary disease including tuberculosis, lung cancer, chronic bronchitis or emphysema
4. History of pneumonia, influenza or whooping cough within the past 30 days.
5. History of asthma that required any treatment within 2 weeks of study
6. T > 38.5oC with no history of anti-pyretic medication for > 24 hours from screening visit
7. History of inhalational exposure (chemical, smoke, water, etc.) within the past 6 months
8. Chest X-ray suggestive of granulomatous disease, malignancy, COPD, bronchiectasis, pneumonia, pleural processes or other underlying pulmonary disease
9. Active, concurrent concomitant disease which might limit the ability of the subject to participate in the study as determined by the Investigator (i.e., diabetes mellitus, congestive heart failure, unstable angina, etc.)
10. Prior or current renal disease; calculated creatinine clearance < 30 ml/min (calculated ClCr < 30)
11. Known immune deficiency condition
12. Use of opioids or anticonvulsants within 3 days of study screening.
13. Known hypersensitivity to memantine or lozenge excipients.
14. Current oral lesions or abnormal findings on buccal examination done at study screening.
15. History of oropharyngeal or gastroesophageal carcinoma, or gastro/esophageal/duodenal resection.
16. Subject has clinically significant abnormal laboratory test results at the screening visit. (Subject may be enrolled by exception, as determined by the Principal Investigator and consented by Cerecor's Medical Monitor.)
17. Any clinically significant finding on the ECG done at the screening visit, as determined by the investigator. (Subject may be enrolled by exception, as determined by the Principal Investigator and consented by Cerecor's Medical Monitor).
18. Female subjects who are pregnant, breast feeding or sexually active without contraception.
19. Subject has donated blood or plasma within the last 45 days.
20. Subject has history of alcohol or drug abuse in past 2 years.
21. Subject has a positive drug screen.
22. Subject has a positive HIV, Hepatitis B or Hepatitis C test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in cough count, active vs placebo treatment period | Daily for 48 hours

SECONDARY OUTCOMES:
Safety | Daily over 3 days
  The evaluation of treatment safety will take into account the recorded adverse events, vital signs, clinical and laboratory assessments and the buccal cavity examination

CONTACTS AND LOCATIONS:
Locations (5):
- Chile (2):
  - Clinica Las Lilas, Santiago
  - Biomedical Research Group, Santiago
- Peru (3):
  - Clinica Internacional Sede Lima, Lima
  - Clinica Internacional Sede San Borja, Lima
  - Unidad de Investigación Clinica San Pablo, Lima